CLINICAL TRIAL: NCT07116252
Title: Effect of Sequential Versus Continous Chelation Protocols on Postoperative Endodontic Pain and Matrix Metalloproteinase-9 Levels: A Randomized Clinical Study
Brief Title: Effect of Different Irrigation Protocols on Postoperative Endodontic Pain and Inflammation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrahman elkholy, Assisstant lecturer of endodontics, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Endodontics
Record Dates: First submitted 2025-07-05; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Irrigation Solution; Postoperative Pain; Inflammation; Endodontic Treatment
Keywords: Clodronate; HEBP; MMP-9; EDTA; Continous chelation
MeSH Terms: conditions — Pain, Postoperative; Inflammation | interventions — Edetic Acid; Etidronic Acid; Clodronic Acid; Sodium Hypochlorite

STUDY DESIGN:
Intervention Model Description: 5 groups with different treatment protocols to assess two parameters
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- 17% EDTA - sequential chelation (Experimental): Irrigation by 2.5% NaOCl during instrumention and a final rinse by 17% EDTA (sequential chelation protocol)
  Interventions: Procedure: EDTA
- 9% HEBP - sequential chelation (Experimental): Irrigation by 2.5% NaOCl during instrumention and a final rinse by 9% HEBP (sequential chelation protocol)
  Interventions: Procedure: Etidronate
- 0.26 M (7.6%) clodronate - sequential chelation (Experimental): Irrigation by 2.5% NaOCl during instrumention and a final rinse by 0.26 M (7.6%) clodronate (sequential chelation protocol)
  Interventions: Procedure: clodronate
- 2.5% NaOCl + 9% HEBP - continous chelation (Experimental): Irrigation by 2.5% NaOCl + 9% HEBP during instrumention and as final rinse (continous chelation protocol)
  Interventions: Procedure: Etidronic acid /sodium hypochlorite
- 2.5% NaOCl + 0.26 M (7.6%) clodronate - continuous chelation (Experimental): Irrigation by 2.5% NaOCl + 0.26 M (7.6%) clodronate during instrumention and as final rinse (continous chelation protocol)
  Interventions: Procedure: clodronate + sodium hypochlorite

INTERVENTIONS:
Procedure: EDTA — 17% EDTA as a final rinse after instrumentaion (sequential chelation)
  Other Names: 17% Ethylenediaminetetraacetic Acid.
  Arms: 17% EDTA - sequential chelation
Procedure: Etidronate — 9% HEBP as a final rinse after instrumentation (sequential chelation)
  Other Names: 9% HEBP or HEDP (1-Hydroxyethylidene-1,1-bisphosphonate)
  Arms: 9% HEBP - sequential chelation
Procedure: clodronate — 0.26 M (7.6%) clodronate as a final rinse after instrumentation (sequential chelation)
  Other Names: 0.26 M (7.6%) clodronate or clodronic acid
  Arms: 0.26 M (7.6%) clodronate - sequential chelation
Procedure: Etidronic acid /sodium hypochlorite — (2.5% NaOCl + 9% HEBP) during instrumentation and as a final rinse after instrumentation (continous chelation)
  Other Names: 2.5% NaOCl + 9% HEBP - continous chelation
  Arms: 2.5% NaOCl + 9% HEBP - continous chelation
Procedure: clodronate + sodium hypochlorite — 2.5% NaOCl + 0.26 M (7.6%) clodronate during instrumentation and as a final rinse after instrumentation (continuous chelation)
  Other Names: 2.5% NaOCl + 0.26 M (7.6%) clodronate - continuous chelation
  Arms: 2.5% NaOCl + 0.26 M (7.6%) clodronate - continuous chelation

SUMMARY:
This study aims to improve the postoperative endodontic outcome by assessing the effect of different irrigants on postoperative endodontic pain and their anti-inflammatory effects.

DETAILED DESCRIPTION:
Alternating application of ethylenediaminetetraacetic acid (EDTA) and sodium hypochlorite (NaOCl) is frequently recommended for removal of organic and inorganic tissues debris including the smear layer. But EDTA can cause loss of available chlorine affecting organic tissue dissolving ability of NaOCl when mixed with it. Etidronic acid is a first-generation bisphosphonate. It is a mild chelator that is compatible with NaOCl in the short term without affecting available chlorine, a concept that has been termed 'continuous chelation'. Clodronate also, was identified with improved stability in NaOCl mixtures compared with EDTA and etidronate.

Aim: Assessment of postoperative endodontic pain and matrix metalloproteinase-9 levels after sequential versus continous chelation protocols.

Methods: This study will be conducted on 75 patients having necrotic pulp with asymptomatic apical periodontitis. Patients will be randomly divided into five groups (Group 1: 2.5% NaOCl during instrumentation then sequential chelation by 17% EDTA, Group 2: 2.5% NaOCl during instrumentation then sequential chelation by 9% HEBP, Group 3: 2.5% NaOCl during instrumentation then sequential chelation by 0.26 M (7.6%) clodronate, Group 4: continuous chelation during instrumentation by 2.5% NaOCl + 9% HEBP, Group 5: continuous chelation by 2.5% NaOCl + 0.26 M (7.6%) clodronate). Postoperative pain will be assessed after 6, 12, 24, 48 hours and 7 days after the first visit using a numerical rating scale. MMP-9 levels in periapical tissues will be quantified using a commercially available ELISA kit applied on the periapical samples that will be collected after the final rinse (S1) and after one week (S2).

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with a single rooted tooth (maxillary anteriors and mandibular premolars) with closed apex and a single patent canal type I in Vertucci's classification (Vertucci et al., 1974)
2. Having a necrotic pulp and asymptomatic apical periodontitis (periapical lesion).
3. Periapical lesions of endodontic origin with a diameter ranging from 2 to 5mm, having a periapical index score of 4 or 5 (Orstavik, Kerekes and Eriksen, 1986)

Exclusion Criteria:

(i) Patients with pain before treatment (ii) Patients having chronic condition requiring the intake of anti-inflammatory/antibiotic drugs.

(iii) Teeth having non-restorable tooth with gross carious lesions, fractures, internal or external root resorption or cracks involving the periodontium.

(iv) Root canals in which patency for periapical fluid sampling could not be achieved.

(v) immune-compromised patients or patients with complicated systemic diseases, physical disability or psychological problems (vi) patients received antibiotic therapy within the last 3months. (vii) Teeth associated with bone expansion or with a history of endodontic treatment.

(viii) Teeth with periodontal pockets deeper than 4mm, with or without concomitant or combined endo-perio communication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain assessment using Numerical Rating Scale NRS | Postoperative pain was assessed after 6, 12, 24, 48 hours and 7 days after the first visit using a numerical rating scale NRS
  Postoperative pain is assessed after 6, 12, 24, 48 hours and 7 days after the first visit using a numerical rating scale NRS where the patient is asked to select the number representing the pain intensity as follow '0' representing no pain and '10' being the worst pain
MMP-9 levels in periapical tissues using periapical fluid samples using a commercially available ELISA kit | After the final rinse (S1) and after one week (S2).
  MMP-9 levels in periapical tissues are quantified using a commercially available ELISA kit applied on the periapical samples that will be collected after the final rinse (S1) and after one week (S2).

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Fayyad, Study Director — Professor of endodontics, faculty of dentistry, Suez Canal University; Dalia Abdallah, Study Director — Associate Professor of endodontics, faculty of dentistry, Suez Canal University
Locations (1):
- Faculty of dentistry, suez canal university, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol and results
Supporting Information: Study Protocol

REFERENCES:
- [Background] La Rosa GRM, Plotino G, Nagendrababu V, Pedulla E. Effectiveness of continuous chelation irrigation protocol in endodontics: a scoping review of laboratory studies. Odontology. 2024 Jan;112(1):1-18. doi: 10.1007/s10266-023-00835-8. Epub 2023 Jul 11. PMID 37433927
- [Background] Rath PP, Yiu CKY, Matinlinna JP, Kishen A, Neelakantan P. The effects of sequential and continuous chelation on dentin. Dent Mater. 2020 Dec;36(12):1655-1665. doi: 10.1016/j.dental.2020.10.010. Epub 2020 Nov 5. PMID 33162115
- [Background] Bassam S, El-Ahmar R, Salloum S, Ayoub S. Endodontic postoperative flare-up: An update. Saudi Dent J. 2021 Nov;33(7):386-394. doi: 10.1016/j.sdentj.2021.05.005. Epub 2021 Jun 3. PMID 34803278
- [Background] Ahmed GM, El-Baz AA, Hashem AA, Shalaan AK. Expression levels of matrix metalloproteinase-9 and gram-negative bacteria in symptomatic and asymptomatic periapical lesions. J Endod. 2013 Apr;39(4):444-8. doi: 10.1016/j.joen.2012.11.009. Epub 2013 Jan 16. PMID 23522533
- [Background] Zollinger A, Mohn D, Zeltner M, Zehnder M. Short-term storage stability of NaOCl solutions when combined with Dual Rinse HEDP. Int Endod J. 2018 Jun;51(6):691-696. doi: 10.1111/iej.12875. Epub 2017 Dec 5. PMID 29121393
- [Background] Wright PP, Cooper C, Kahler B, Walsh LJ. From an assessment of multiple chelators, clodronate has potential for use in continuous chelation. Int Endod J. 2020 Jan;53(1):122-134. doi: 10.1111/iej.13213. Epub 2019 Sep 26. PMID 31483863
- [Background] Ballal NV, Gandhi P, Shenoy PA, Shenoy Belle V, Bhat V, Rechenberg DK, Zehnder M. Safety assessment of an etidronate in a sodium hypochlorite solution: randomized double-blind trial. Int Endod J. 2019 Sep;52(9):1274-1282. doi: 10.1111/iej.13129. Epub 2019 May 13. PMID 30993696